CLINICAL TRIAL: NCT06221332
Title: The Effect of Sacral Erector Spinae Plane Block on the Quality of Recovery After Vaginal Birth: A Double-blind Prospective Randomized Controlled Study.
Brief Title: Sacral Erector Spinae Plane Block in Normal Birth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Muhammed Halit Satici, Specialist, M.D., Department of members Anesthesiology and Reanimation, Konya City Hospital, M.D, Konya City Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: vaginal birth
Record Dates: First submitted 2023-12-27; First posted 2024-01-24 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SACRAL EREKTÖR SPİNAE PLANE BLOK (Active Comparator): Pregnant women in Group S will be given 10 cc bupivacaine solution of 0.25% bupivacaine on both sides.
  Interventions: Other: % 0.25 bupivakain 20cc
- control group (Active Comparator): Pregnant women in Group K will be injected with 10 cc of saline on both sides.
  Interventions: Other: 20 cc saline

INTERVENTIONS:
Other: % 0.25 bupivakain 20cc — Pregnant women in group S will be given 0.25% bupivacaine, 10 cc on each side.
  Arms: SACRAL EREKTÖR SPİNAE PLANE BLOK
Other: 20 cc saline — Pregnant women in Group K will be given 10 cc of saline on both sides.
  Arms: control group

SUMMARY:
Pregnant women feel severe pain during normal birth and in the postpartum period. Preventing pain during and after birth is very important for both the mother and the baby. Rapid recovery in the postoperative period in pregnant women is very important for both mother and baby. To evaluate this recovery, the quality of recovery-10 scores developed by Shalev et al. are used in pregnant women. Our study will be the first in the literature to use sacral erectör spinae plane block (S-ESPB) in normal birth. Our primary aim in this study is to evaluate the effects of S-ESPB on the quality of recovery and recovery at the 24th hour in pregnant women who will undergo vaginal birth with epidural analgesia, using the Quality of Recovery-10T scores.

DETAILED DESCRIPTION:
Pregnant women feel severe pain during normal birth and in the postpartum period. Preventing pain during and after birth is very important for both the mother and the baby. Rapid recovery in the postoperative period in pregnant women is very important for both mother and baby. To evaluate this recovery, the quality of recovery-10 scores developed by Shalev et al. are used in pregnant women. Our study will be the first in the literature to use sacral erectör spinae plane block in normal birth. Our primary aim in this study is to evaluate the effects of sacral erectör spinae plane block on the quality of recovery and recovery at the 24th hour in pregnant women who will undergo vaginal birth with epidural analgesia, using the Quality of recovery-10T score. the numeric rating scale at the 0-15th minute-30th minute-45th minute-1-2-4-8-12-24th hour after the S-ESPB application, and to evaluate the patient satisfaction at the 24th hour with a Likert scale. , the total amount of rescue analgesic ( bupivacaine ) consumed since the application of sacral erectör spinae plane block, the number of pregnant women given oxytocin, the time of the first breastfeeding, complications in the mother (fever, nausea, vomiting, motor block, hip pain), the need for antiemetics, the baby's 1st and 5th minutes. Apgar score at the 1st-2nd-3rd week of birth. is to evaluate the duration of the phases .

ELIGIBILITY:
Inclusion Criteria:

* 36-42. Pregnant women who are their gestational age and request epidural anesthesia
* Pregnant women aged 18-42 with ASA II
* Pregnant women who will stay in the hospital for at least 24 hours
* Primiparous pregnant women who will have a planned normal birth
* Singleton births with vertex presentation

Exclusion Criteria:

* Pregnant women who do not want to give consent
* Regional anesthesia is contraindicated
* Pregnant women who use anticoagulants and have an abnormal bleeding profile
* Pregnant women with infection in the area to be treated
* Emergency cases and pregnant women who had a birth with instruments (forceps and vacuum)

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women who will have normal birth
Enrollment: 40 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Quality of recovery (10T) scores | One day
  The primary evaluation criterion will be the recording of Quality of Recovery-10T scores, which indicate the quality of recovery of pregnant women at the 24th hour after birth. Quality of Recovery-10T ( Minumum: 0 = Very bad, Maximum: 100= Perfect).

CONTACTS AND LOCATIONS:
Overall Officials: MUHAMMED H SATICI, M.D., Principal Investigator — Konya City Hospital
Locations (1):
- Konya City Hospital, Konya, Turkey (Türkiye)